CLINICAL TRIAL: NCT01875536
Title: Efficacy of Coupling Repetitive Transcranial Magnetic Stimulation and Conventional Physical Therapy to Reduce Upper Limb Spasticity in Stroke Patients
Brief Title: rTMS and Conventional Physical Therapy After Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Professor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rTMS_Physical Therapy_stroke
Record Dates: First submitted 2013-06-06; First posted 2013-06-12 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Stroke
Keywords: transcranial magnetic stimulation; spasticity; physiotherapy; Rehabilitation
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rTMS (Experimental): The experimental group received rTMS to the primary motor cortex of the unaffected side in 10 sessions, 3 days per week, and conventional physical therapy
  Interventions: Device: rTMS; Behavioral: conventional physical therapy
- control (Sham Comparator): The control group received sham stimulation (same area as the experimental group) in 10 sessions, 3 days per week, and conventional physical therapy
  Interventions: Behavioral: conventional physical therapy

INTERVENTIONS:
Device: rTMS — The subjects were seated in a comfortable chair with head and arm rests. Focal TMS of the motor cortex was performed with a 70-mm figure-8 coil attached to magnetic stimulator stimulation parameters : frequency of 1Hz on the uninjured hemisphere by stroke; 1500 pulses with an intensity of 90% of MT 10 sessions of rTMS, one per day, always before conventional physical therapy
  Arms: rTMS
Behavioral: conventional physical therapy — The physical therapy program was composed of the activities of flexibility, transfer and posture, strength, coordination, balance, and sensory stimulation. The physical therapy was applied for about 30 minutes, three days per week.

SUMMARY:
Given previous evidence that non invasive brain stimulation enhances the effects of conventional therapies, this randomized sham-controlled trial with 4-weeks follow-up aimed to determine if the repetitive transcranial magnetic stimulation (rTMS)combined with conventional physical therapy (VRT) would be superior to physical therapy in improving upper limb function and quality of life with chronic stroke individuals.

ELIGIBILITY:
Inclusion Criteria:

* stroke onset ≥ 6 months;
* muscle tone at the wrist with a modified Ashworth scale (MAS) score between 1+ and 3;
* minimum age of 30 years old and maximum age of 75 years;
* absence of cognitive impairment, as determined by the cut-off scores on the Mini-mental state exam

Exclusion Criteria:

* history of seizure or cerebral aneurism;
* antispasticity drugs within 6 months before enrollment;
* previous surgery involving metallic implants;
* unstable vital signs;
* other neurological diseases
* aphasia

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from Modified Ashworth scale | at baseline, 1 month and 2 months
  Modified Ashworth scale (MAS) uses a 6-point scale to score the average resistance to passive movement for each joint. In this study, the tonus of the wrist flexor muscles was tested
change from spinal excitability via Hoffmann reflex of the median nerve | at baseline, 1 month and 2 months
  assess the effects of the intervention (rTMS and physical therapy) on spinal excitability as measured by the change The Hmax/Mmax ratio (calculated by dividing the maximal amplitude of the H wave by that of the M wave in median nerve) before (baseline), after treatment and after follow-up

SECONDARY OUTCOMES:
change from Fugl-Meyer assessment | at baseline, 1 month and 2 months
  The Fugl-Meyer assessment (FMA) is considered the gold standard for evaluating the motor function recovery. It is designed to assess motor functioning, balance, sensation, and joint functioning. It is applied within clinical and in research contexts to determine the disease severity, describe motor recovery, and plan and assess interventions. In the present study, the 33-item of the UL section was employed. The items are rated on 3-point ordinal scale, as follows: 0= unable to perform; 1= partial ability to perform; and 2= near normal ability to perform. The UL subscale evaluates motor function recovery in six domains: flexor and extensor synergies, non-synergic movements, wrist and hand movements, and coordination and speed
change from cortical excitability via single transcranial magnetic stimulation | per-session: at baseline and one hour (after physical therapy)
  assess the effects of the intervention (rTMS and physical therapy) on motor cortex excitability as measured by the change in motor evoked potential (using transcranial magnetic stimulation) before and after each session

OTHER OUTCOMES:
change from stroke specific quality of life scale | at baseline, 1 month and 2 months
  the stroke specific quality of life scale (SSQOL) is used to provide an assessment of health-related quality of life specific to patients with stroke. The scale is a self-report (reference to the past two weeks) containing 49 items distributed into 12 domains (mobility, energy, upper extremity function, work/productivity, mood, self-care, social roles, family roles, vision, language, thinking and personality), rated on a 5-point scale. The total score (maximum 245) and the upper extremity function scores (maximum of 25) can be considered for analyses. The Brazilian version of the SSQOL was used in this study

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Neuroscience Laboratory-LANA, Recife, Pernambuco, Brazil